CLINICAL TRIAL: NCT00763009
Title: Persantine: Variation in Response Trial
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Limited numbers of patients qualified for trial
Sponsor: UConn Health (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 02-202-1; A-13147.1
Record Dates: First submitted 2008-09-24; First posted 2008-09-30 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Dipyridamole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All subjects receive dipyridamole (Other): Compare to baseline
  Interventions: Drug: dipyridamole

INTERVENTIONS:
Drug: dipyridamole — 0.28mg/kg over 4 minutes intravenously x three doses; totalling 0.84mg/kg intravenously
  Other Names: Persantine

SUMMARY:
The primary objective of this study is to understand why different people respond differently to the medication Persantine. The effects of Persantine will be evaluated by performing echocardiograms, blood tests and by measuring the flow of blood in the arteries of the heart in patients undergoing a clinically indicated percutaneous coronary intervention.

DETAILED DESCRIPTION:
Participants will receive three doses of Persantine intravenously for the research study. Before and after receiving the Persantine doses, patients will have an echocardiogram and coronary artery blood flow will be measured. Blood tests,measure the function of the adenosine transporter. In addition variations in the gene for the adenosine transporter will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 21 years old
* Patient undergoing cardiac catheterization with planned PTCA or with a significant coronary lesion of either the LAD or Circumflex

Exclusion Criteria:

* Theophylline or oral Persantine use in 24hrs
* Second or third degree AV block, or sick sinus syndrome without a functioning pacemaker
* Active asthma or bronchospasm
* Patients with severe hepatic insufficiency
* Patients experiencing an acute transmural infarction at the time of the index visit
* Conditions that are known to affect resistive vessel function or myocardial flow

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2002-09 (Actual); Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Azrin, MD, Principal Investigator — University of Connecticut; Bruce T Liang, MD, Study Chair — University of Connecticut
Locations (1):
- UCONN Health Center, Farmington, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study terminated due to difficulty enrolling
Pre-assignment Details: Study terminated due to difficulty enrolling
Groups:
- All Subjects Receive Dipyridamole: There is only a single arm
  dipyridamole: 0.28mg/kg over 4 minutes intravenously x three doses; totalling 0.84mg/kg intravenously
Period: Overall Study
Arm/Group | All Subjects Receive Dipyridamole
Started | 8
Completed | 7
Not Completed | 1
Not completed — Coronary Anatomy unsuitable | 1

BASELINE CHARACTERISTICS:
Groups:
- Dipyridamole: Pre: Baseline Results prior to administration of Dipyridamole. Post: Results post adminsitration of Dipyridamole
Arm/Group | Dipyridamole
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: To Determine if There is a Subgroup of Patients That Have an Abnormal Adenosine Transporter Expression, or Abnormal Adenosine Transporter Protein Function.
Description: To determine if there is a subgroup of patients that have an abnormal adenosine transporter expression, or abnormal adenosine transporter protein function. All were responsive Study terminated due to difficulty enrolling
Time Frame: 6-12 months
Population: All patients responded. Function and Expression of the Transporter were therefore not performed.
  The study was terminated due to poor enrollment
Arm/Group | All Subjects Receive Dipyridamole
Number analyzed (Participants) | 0

2. Secondary Outcome: To Determine the Clinical Significance of Variations in Adenosine Transfer Function on Coronary Flow.
Time Frame: 6-12 months
Population: The study was terminated due to poor enrollment
Arm/Group | All Subjects Receive Dipyridamole
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | All Subjects Receive Dipyridamole
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
Trial terminated early due to poor patient enrollment. All patients responded hemodynamically. Therefore, analysis of responders vs non-responders could not be performed. Adenosine transporter was not analyzed since there was no comparator group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No